CLINICAL TRIAL: NCT03121820
Title: A Two-way Crossover, Open-label, Single-dose, Fasting, Bioequivalence Study of Memantinol® (JSC "GEROPHARM", Russia) 20 mg Tablets Versus Akatinol Memantine® (Merz Pharma GmbH & Co. KGaA, Germany) 20 mg Tablets in Normal Healthy Subjects
Brief Title: Fasting Bioequivalence Study of Memantinol 20 mg Tablets Versus Akatinol Memantine® 20 mg Tablets In Normal Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Geropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BIOMEM-20
Record Dates: First submitted 2017-04-18; First posted 2017-04-20 (Actual); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2017-07

CONDITIONS: Bioequivalence, AUC, Cmax, Pharmacokinetics
MeSH Terms: interventions — Memantine

STUDY DESIGN:
Intervention Model Description: two-way crossover
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Memantinol tablets, 20 mg (Experimental): Treatment A: a single oral dose of memantin 20 mg film-coated tablet (JSC "GEROPHARM", Russia - test)
  Interventions: Drug: Memantinol tablets, 20 mg
- Akatinol Memantine® tablets, 20 mg (Active Comparator): Treatment B: a single oral dose of memantin 20 mg film-coated tablet (Merz Pharma GmbH & Co. KGaA, Germany - reference)
  Interventions: Drug: Akatinol Memantine® tablets, 20 mg

INTERVENTIONS:
Drug: Memantinol tablets, 20 mg — Bioequivalence Memantine Hydrochloride (JSC "GEROPHARM", Russia) 20 mg film-coated tablets fasting condition
  Other Names: memantine
  Arms: Memantinol tablets, 20 mg
Drug: Akatinol Memantine® tablets, 20 mg — Bioequivalence Memantine Hydrochloride (Merz Pharma GmbH & Co. KGaA, Germany) 20 mg film-coated tablets fasting condition
  Other Names: memantine
  Arms: Akatinol Memantine® tablets, 20 mg

SUMMARY:
This study are two-way crossover, open-label, single-dose, fasting, bioequivalence study of Memantinol® (JSC "GEROPHARM", Russia) 20 mg tablets versus Akatinol Memantine® (Merz Pharma GmbH & Co. KGaA, Germany) 20 mg tablets in normal healthy subjects

DETAILED DESCRIPTION:
Study to evaluate the bioequivalence of orally administered memantinol preparations, film-coated tablets, 20 mg

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Healthy male and female subjects aged 18 to 45 years.
* Verified diagnosis is "healthy" according to data Standard clinical, laboratory and Instrumental methods of examination.
* Have a body mass index between 18,5 and 27 kg/m2.
* Females must have a negative pregnancy test.
* Subjects must use, with their partner, methods of highly effective contraception; if the Hormonal contraceptives was used they must canceled have at least 2 month before the study.

from the time of IMP administration until 3 months after the last dose of IMP.

Exclusion Criteria:

* History of serious allergic problems/events
* Medicinal intolerance.
* History of allergic reactions to memantine or investigator's product components
* Any acute and chronic diseases of the cardiovascular system, cardiovascular, bronchopulmonary, neuroendocrinal systems, as well as diseases of the gastrointestinal tract, liver, kidneys, blood.
* Acute infectious diseases in less than 4 weeks before the start of the study.
* Subjects who have taken medication 4 weeks preceding before the study.
* Subjects who have taken any drugs known effects on hemodynamics or to induce or inhibit hepatic drug metabolism within 30 days prior to administration of the study medication (examples of inducers: barbiturates, omeprazole, etc.).
* Donation of plasma (450 mL or more) within 2 month prior to administration of the study medication.
* History of significant alcohol or drugs abuse or any indication of the regular use of more than 10 units of alcohol per week (1 Unit = 200 mL of wine or 500 mL of beer or 50 mL of alcohol 40%).
* Smokers.
* Participation in other clinical training is less than than for 3 months before the study.
* Lack of signed informed consent form.
* ECG or vital signs abnormalities (clinically significant).
* Positive testing for alcohol, drugs, pregnancy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2016-11-19 (Actual); Study Completion 2016-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Igor Makarenko, MD, PhD, Study Chair — Igor.Makarenko@geropharm.com
Locations (1):
- City Clinical Hospital № 15 named. O.M.filatova, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited at GKB № 15 im. O. M. Filatova Public Healthcare Institution of Department of health care of Moscow, Russian Federation between October and November 2016
Pre-assignment Details: 18 participants recruited; 25 screened, 7 excluded (5 did not meet inclusion criteria and 2 refused participation).
Groups:
- Memantinol First, Then Akatinol Memantine®: First Intervention Period (3 day):
  Memantinol tablet: Single administered dose of Memantinol ( 20 mg memantin) in a fasting state
  (21 day washout period)
  Second Intervention Period (3 day):
  Akatinol Memantine® tablet: Single administered dose of Memantinol ( 20 mg memantin) in a fasting state
- Akatinol Memantine® First, Then Memantinol: First Intervention Period (3 day):
  Akatinol Memantine® tablet: Single administered dose of Memantinol ( 20 mg memantin) in a fasting state
  (21 day washout period)
  Second Intervention Period (3 day):
  Memantinol tablet: Single administered dose of Memantinol ( 20 mg memantin) in a fasting state
Period: First Period
Arm/Group | Memantinol First, Then Akatinol Memantine® | Akatinol Memantine® First, Then Memantinol
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Second Period (After Washout)
Arm/Group | Memantinol First, Then Akatinol Memantine® | Akatinol Memantine® First, Then Memantinol
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantinol First, Then Akatinol Memantine® | Akatinol Memantine® First, Then Memantinol | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of Memantinol by Assessment of Area Under the Curve From Time Zero Extrapolated to Infinity (AUC(0-inf))
Description: Comparison of the pharmacokinetic profile in terms of plasma concentration-time curve from time zero extrapolated to infinity, AUC(0-inf), of memantinol sourced in Memantinol® (JSC "GEROPHARM", Russia) and Akatinol Memantine® (Merz Pharma GmbH & Co. KGaA, Germany)
Time Frame: 0 hours (pre-dose), as well as at 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 9, 10, 12, 16, 24, 36, 48 and 72 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Memantinol Tablets, 20 mg | Akatinol Memantine® Tablets, 20 mg
Number analyzed (Participants) | 18 | 18
ng*h/mL | 1920.362 (449.289) | 2096.669 (537.147)
Statistical Analysis 1: Comparison: Memantinol Tablets, 20 mg vs Akatinol Memantine® Tablets, 20 mg; Memantinol 20 mg Tablets Versus Akatinol Memantine® 20 mg; Test type: Non-Inferiority or Equivalence — The analysis was conducted using an analysis of variance (ANOVA) including fixed effects for treatment, sequence, period and subject within sequence. All pharmacokinetic parameters were log-transformed prior to analysis. Bioequivalence was concluded, when the 90% confidence interval (CI) for the geometric mean ratios were fully contained within the predefined equivalence limits of 80.00 % to 125.00 %; p = 0.05, Test/Ref Geometric mean ratio x 100; Bioequivalence is established when 90% Confidence Interval falls within 80.00 % -125.00 %; Test/Ref Geometric mean ratio x 100 = 93.8, 90% CI 2-sided [88.25 to 99.77]

2. Primary Outcome: Pharmacokinetics of Memantinol by Assessment of Observed Maximum Plasma Concentration (Cmax)
Description: Comparison of the pharmacokinetic profile in terms of observed maximum plasma concentration, taken directly from the individual concentration-time curve, Cmax, of memantinol sourced in Memantinol® (JSC "GEROPHARM", Russia) and Akatinol Memantine® (Merz Pharma GmbH & Co. KGaA, Germany)
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Memantinol Tablets, 20 mg | Akatinol Memantine® Tablets, 20 mg
Number analyzed (Participants) | 18 | 18
ng/mL | 34.617 (8.302) | 37.578 (8.858)
Statistical Analysis 1: Comparison: Memantinol Tablets, 20 mg vs Akatinol Memantine® Tablets, 20 mg; Memantinol 20 mg Tablets Versus Akatinol Memantine® 20 mg; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.05, Test/Ref Geometric mean ratio x 100; Bioequivalence is established when 90% Confidence Interval falls within 80.00 % -125.00 %; Test/Ref Geometric mean ratio x 100 = 92.3, 90% CI 2-sided [86.37 to 98.55]

ADVERSE EVENTS:
Groups:
- Memantinol Tablets, 20 mg: Active experimental drug
  Memantinol: Single orally administered dose of Memantinol (20 mg memantine) in a fasting state
- Akatinol Memantine® Tablets, 20 mg: Active comparator
  Akatinol Memantine®: Single orally administered dose of Akatinol Memantine® (20 mg memantine) in a fasting state
Arm/Group | Memantinol Tablets, 20 mg | Akatinol Memantine® Tablets, 20 mg
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 2/18 | 2/18
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Memantinol Tablets, 20 mg (N=18) | Akatinol Memantine® Tablets, 20 mg (N=18)
Dizziness (Nervous system disorders) | 2 | 2 — The volunteers during period, 2.5 hours after taking the test drug (20 mg orally) was dizzy. Deviations in any Analyzed indicators were not revealed. There was no volunteer Action taken. AE resolved full recovery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a publication (e.g., in a scientific journal) based on the results of this study is envisaged, approval from GEROPHARM will be obtained and a draft manuscript will be submitted to GEROPHARM for scrutiny and comment. The choice of conduit will be mutually agreed on by the Principal Investigator and GEROPHARM.